CLINICAL TRIAL: NCT00828919
Title: CONTINUING ACCESS TO THE TYROSINE KINASE INHIBITOR OF VEGFR-2, AG-013736 (A406) FOR PATIENTS PREVIOUSLY RECEIVING AG-013736 IN CLINICAL TRIALS
Brief Title: Continuing Access to Axitinib (A406- AG- 013736 ) For Patients Previously Receiving AG 013736 In Clinical Trials
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Masking: None | Purpose: Treatment
Other Study IDs: A4061008; 2005-000051-15 (EudraCT Number)
Record Dates: First submitted 2009-01-23; First posted 2009-01-26 (Estimated); Results first posted 2024-12-03 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Solid Tumors
Keywords: VEGFR inhibitor; angi-angiogenic; tyrosine kinase inhibitor
MeSH Terms: interventions — Axitinib; Crizotinib

STUDY DESIGN:
Intervention Model Description: This is a continuing access, open label study for patients to receive monotherapy or combination therapy based on previous treatment received in parent protocol
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (Experimental): Patients continue the same treatment (axitinib monotherapy or in combination with crizotinib) as in prior axitinib study
  Interventions: Drug: axitinib; Drug: crizotinib

INTERVENTIONS:
Drug: axitinib — BID oral tablets. dose of axitinib (AG 013736) will be the same as they were taking in the previous trial
  Other Names: AG-013736
Drug: crizotinib — BID oral Capsules. Dose of crizotinib will be the same taken in previous axitinib trial.
  Other Names: PF-02341066

SUMMARY:
To allow continuation of axitinib (AG 013736) treatment to patients experiencing clinical benefit in a closing axitinib trial

DETAILED DESCRIPTION:
This is a roll over study aimed to provide continued access to axitinib (monotherapy or combination, according to treatment received in prior axitinib study) to patients who have documented stable, or responding disease, or received clinical benefit (as defined by protocol) at the time of the prior study closure.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were assigned to an axitinib (AG-013736) containing treatment arm in a previous clinical trial
* Patients who were receiving axitinib (AG-013736) tablets at the time their previous trial ended
* Patients who have stable (SD) or responding disease (PR or CR) documented by the appropriate radiological, clinical, or laboratory assessments within 12 weeks before enrollment (Note: response criteria from the previous axitinib (AG-013736) protocol should be used to determine stable or responding disease).
* Patients who have progressive disease (PD) but have experienced "clinical benefit" as defined in the study protocol

Exclusion Criteria:

* Patients may not participate in this trial if the conditions for continuing treatment in the previous axitinib (AG-013736) protocol are not met

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2003-03-07 (Actual); Primary Completion 2023-08-14 (Actual); Study Completion 2023-08-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (33):
- United States (17):
  - UC Irvine Medical Center, Orange, California
  - University of California Irvine Medical Center - Chao Family Comprehensive Cancer Center, Orange, California
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - UCLA Hematology-Oncology-Santa Monica, Santa Monica, California
  - University of Chicago Hospitals, Chicago, Illinois
  - Johns Hopkins University, Baltimore, Maryland
  - Johns Hopkins Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland
  - University of Michigan Health System, Ann Arbor, Michigan
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - The Cleveland Clinic, Cleveland, Ohio
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - The University of Texas M.D. Anderson Cancer Center, Houston, Texas
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - Providence Regional Medical Center Everett - Providence Regional Cancer Partnership, Everett, Washington
  - Providence Regional Medical Center Everett, Everett, Washington
  - University of Wisconsin - Hospital and Clinics, Madison, Wisconsin
- Czechia (2):
  - Fakultni nemocnice Olomouc, Olomouc, Czech Republic
  - Nemocnice Na Bulovce, Prague
- Hopital de la Pitie Salpetriere, Paris, France
- Charité - Universitaetsmedizin Berlin, Charité Campus Mitte, Berlin, Germany
- Semmelweis Egyetem Altalanos Orvostudomanyi Kar, Budapest, Hungary
- Italy (2):
  - Fondazione IRCCS, Istituto Nazionale Tumori, Laboratorio, Milan
  - Fondazione IRCCS, Istituto Nazionale Tumori, S.S.D Oncologia Medica dei Tumori testa-collo, Milan
- Japan (5):
  - National Cancer Center Hospital East, Kashiwa, Chiba
  - Kinki University Hospital, Sayama, Osaka
  - Chiba Cancer Center, Chiba
  - Kyushu University Hospital, Fukuoka
  - Nagasaki University Hospital, Nagasaki
- FSBSI "N.N. Blokhin Russian Cancer Research Center", Moscow, Russian Federation, Russia
- Samsung Medical Center, Seoul, South Korea
- Taichung Veterans General Hospital, Taichung, Taiwan
- Nottingham City Hospital / Oncology Department, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A4061008&StudyName=Continuing%20Access%20To%20AG-%20013736%20%28A406%29%20For%20Patients%20Previously%20Receiving%20AG%20013736%20In%20Clinical%20Trials

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 52 participants were enrolled in this study, out of which 49 were treated. Enrollment for this study was planned to be conducted into two groups: Axitinib monotherapy and Axitinib combination therapy. However, no participant enrolled in Axitinib combination therapy group.
Pre-assignment Details: Participants receiving axitinib in previous trials began this study with the last dose taken in the parent study. Participants continued to access axitinib on this study as long as there was documented stable disease, responding disease, or clinical benefit at the time of prior study closure.
Groups:
- Axitinib 2 mg: Participants received Axitinib 1 micrograms (mg) twice daily orally.
- Axitinib 3 mg: Participants received Axitinib 1 mg twice daily.
- Axitinib 5 mg: Participants received Axitinib 5 mg twice daily.
- Axitinib 7 mg: Participants received Axitinib 5 mg plus Axitinib 1 mg twice daily.
- Other: Participants who received Axitinib twice daily orally as dose other than 2 mg, 3 mg, 5 mg and 7 mg.
Period: Overall Study
Arm/Group | Axitinib 2 mg | Axitinib 3 mg | Axitinib 5 mg | Axitinib 7 mg | Other
Started | 7 | 9 | 20 | 2 | 11
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 7 | 9 | 20 | 2 | 11
Not completed — Death | 0 | 1 | 2 | 0 | 0
Not completed — Adverse Event | 2 | 2 | 2 | 1 | 3
Not completed — Objective progression or relapse | 4 | 4 | 11 | 0 | 5
Not completed — No longer willing to participate in study | 0 | 0 | 2 | 0 | 0
Not completed — Insufficient Clinical Response | 0 | 1 | 2 | 0 | 0
Not completed — Subject refused continued treatment for reason other than adverse event | 0 | 0 | 0 | 0 | 3
Not completed — Other | 1 | 0 | 1 | 1 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who received at least one dose of axitinib under A4061008 protocol.
Groups:
- Total: Total of all reporting groups
Arm/Group | Axitinib 2 mg | Axitinib 3 mg | Axitinib 5 mg | Axitinib 7 mg | Other | Total
Number analyzed (Participants) | 7 | 9 | 20 | 2 | 11 | 49
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.6 (14.7) | 57.1 (11.3) | 58.5 (4.2) | 68.5 (3.5) | 64.6 (8.6) | 60.4 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4 | 1 | 5 | 14
  Male | 5 | 7 | 16 | 1 | 6 | 35
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 5 | 2 | 4 | 0 | 0 | 11
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 0 | 0 | 1
  White | 2 | 5 | 14 | 2 | 9 | 32
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 2 | 0 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs), Serious TEAEs, Treatment Related TEAEs and Treatment Related Serious TEAEs
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between first dose of study drug and up to 28 days after last dose that were absent before treatment or that worsened relative to pretreatment state. Relatedness of an AE to study drug was based on investigator's assessment. AEs included both serious and non-serious AEs.
Time Frame: Day 1 up to 28 days after last dose of study drug (maximum treatment exposure was 119.56 months; maximum follow-up to approximately 120.56 months)
Population: Safety population included all participants who received at least 1 dose of Axitinib under A4061008 protocol.
Measure: Count of Participants; unit: Participants
Groups:
- Overall: Participants received oral dose of Axitinib (any dose) alone twice daily as they were taking in the previous trial.
Arm/Group | Overall | Axitinib 2 mg | Axitinib 3 mg | Axitinib 5 mg | Axitinib 7 mg | Other
Number analyzed (Participants) | 49 | 7 | 9 | 20 | 2 | 11
Participants
  TEAEs | 49 | 7 | 9 | 20 | 2 | 11
  Serious TEAEs | 21 | 4 | 8 | 5 | 0 | 4
  Treatment Related TEAEs | 47 | 7 | 9 | 18 | 2 | 11
  Treatment Related Serious TEAEs | 15 | 2 | 7 | 3 | 0 | 3

ADVERSE EVENTS:
Time Frame: Day 1 up to 28 days after last dose of study drug (maximum treatment exposure was 119.56 months; maximum follow up to approximately 120.56 months)
Description: Same event may appear as both non-SAE and SAE but what is presented are distinct events. An event may be categorised as serious in one participant and nonserious in another participant or one participant may have experienced both serious and non-serious event. Safety population included all participants who received at least 1 dose of Axitinib under A4061008 protocol.
Arm/Group | Overall | Axitinib 2 mg | Axitinib 3 mg | Axitinib 5 mg | Axitinib 7 mg | Other
All-Cause Mortality (participants affected / at risk) | 5/49 | 1/7 | 1/9 | 3/20 | 0/2 | 0/11
Serious Adverse Events (participants affected / at risk) | 21/49 | 4/7 | 8/9 | 5/20 | 0/2 | 4/11
Other Adverse Events (participants affected / at risk) | 48/49 | 7/7 | 9/9 | 19/20 | 2/2 | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Overall (N=49) | Axitinib 2 mg (N=7) | Axitinib 3 mg (N=9) | Axitinib 5 mg (N=20) | Axitinib 7 mg (N=2) | Other (N=11)
Neutropenia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 0 | 0 | 0
Acute coronary syndrome (Cardiac disorders) | 2 | 0 | 2 | 0 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 3 | 1 | 1 | 1 | 0 | 0
Arrhythmia (Cardiac disorders) | 1 | 0 | 1 | 0 | 0 | 0
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0 | 1 | 0 | 0 | 0
Intracardiac thrombus (Cardiac disorders) | 1 | 0 | 1 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 6 | 0 | 5 | 0 | 0 | 1
Retinal vein occlusion (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 1
Ascites (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 1
Colitis (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 0 | 1 | 1 | 0 | 0
Enterocolitis (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0 | 2 | 0 | 0 | 0
Chest pain (General disorders) | 1 | 0 | 1 | 0 | 0 | 0
Disease progression (General disorders) | 1 | 0 | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 0 | 1 | 0 | 0
Biliary obstruction (Hepatobiliary disorders) | 1 | 0 | 1 | 0 | 0 | 0
Septic shock (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 1 | 0 | 1 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 3 | 0 | 2 | 1 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 0 | 1 | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 0 | 0
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0 | 0 | 0
Lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 1
Aphasia (Nervous system disorders) | 1 | 0 | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 0
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 1 | 0 | 0 | 1 | 0 | 0
Transient global amnesia (Nervous system disorders) | 1 | 0 | 1 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 1 | 0 | 0 | 1 | 0 | 0
Proteinuria (Renal and urinary disorders) | 1 | 1 | 0 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 1 | 0 | 0 | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0 | 0
Pulmonary toxicity (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0 | 0
Cholecystectomy (Surgical and medical procedures) | 1 | 0 | 0 | 1 | 0 | 0
Hypotension (Vascular disorders) | 1 | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Overall (N=49) | Axitinib 2 mg (N=7) | Axitinib 3 mg (N=9) | Axitinib 5 mg (N=20) | Axitinib 7 mg (N=2) | Other (N=11)
Anaemia (Blood and lymphatic system disorders) | 3 | 0 | 0 | 3 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 4 | 0 | 1 | 1 | 0 | 2
Hypothyroidism (Endocrine disorders) | 16 | 3 | 4 | 5 | 1 | 3
Abdominal pain (Gastrointestinal disorders) | 4 | 0 | 1 | 1 | 0 | 2
Abdominal pain upper (Gastrointestinal disorders) | 4 | 0 | 1 | 2 | 0 | 1
Constipation (Gastrointestinal disorders) | 6 | 0 | 2 | 1 | 1 | 2
Diarrhoea (Gastrointestinal disorders) | 30 | 3 | 9 | 10 | 2 | 6
Dyspepsia (Gastrointestinal disorders) | 7 | 0 | 3 | 2 | 0 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 | 1 | 1 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 11 | 1 | 3 | 2 | 2 | 3
Stomatitis (Gastrointestinal disorders) | 3 | 0 | 1 | 2 | 0 | 0
Vomiting (Gastrointestinal disorders) | 4 | 0 | 2 | 2 | 0 | 0
Asthenia (General disorders) | 3 | 0 | 2 | 1 | 0 | 0
Chest pain (General disorders) | 6 | 0 | 3 | 3 | 0 | 0
Chills (General disorders) | 4 | 0 | 1 | 2 | 0 | 1
Fatigue (General disorders) | 21 | 1 | 6 | 6 | 2 | 6
Influenza like illness (General disorders) | 3 | 1 | 2 | 0 | 0 | 0
Oedema (General disorders) | 4 | 1 | 2 | 0 | 0 | 1
Oedema peripheral (General disorders) | 7 | 0 | 3 | 1 | 0 | 3
Pyrexia (General disorders) | 4 | 0 | 2 | 2 | 0 | 0
Nasopharyngitis (Infections and infestations) | 3 | 0 | 1 | 1 | 1 | 0
Rhinitis (Infections and infestations) | 5 | 0 | 2 | 3 | 0 | 0
Sinusitis (Infections and infestations) | 6 | 0 | 2 | 1 | 0 | 3
Tooth infection (Infections and infestations) | 3 | 1 | 2 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 9 | 2 | 3 | 1 | 0 | 3
Urinary tract infection (Infections and infestations) | 3 | 0 | 1 | 0 | 0 | 2
Blood cholesterol increased (Investigations) | 3 | 0 | 0 | 0 | 1 | 2
Blood creatinine increased (Investigations) | 3 | 1 | 1 | 0 | 1 | 0
Weight decreased (Investigations) | 17 | 1 | 5 | 7 | 1 | 3
Decreased appetite (Metabolism and nutrition disorders) | 8 | 2 | 3 | 0 | 1 | 2
Dehydration (Metabolism and nutrition disorders) | 4 | 0 | 2 | 2 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 6 | 0 | 1 | 3 | 1 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 4 | 2 | 1 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 11 | 3 | 2 | 4 | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 0 | 1 | 2 | 1 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 3 | 1 | 0 | 2 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 6 | 1 | 2 | 2 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 9 | 1 | 3 | 3 | 0 | 2
Dizziness (Nervous system disorders) | 6 | 1 | 2 | 1 | 0 | 2
Headache (Nervous system disorders) | 12 | 2 | 3 | 4 | 1 | 2
Paraesthesia (Nervous system disorders) | 4 | 1 | 1 | 1 | 1 | 0
Taste disorder (Nervous system disorders) | 3 | 1 | 1 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 5 | 0 | 1 | 4 | 0 | 0
Dysuria (Renal and urinary disorders) | 4 | 0 | 0 | 2 | 1 | 1
Proteinuria (Renal and urinary disorders) | 14 | 5 | 1 | 5 | 0 | 3
Erectile dysfunction (Reproductive system and breast disorders) | 4 | 0 | 0 | 3 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 8 | 1 | 0 | 4 | 1 | 2
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 9 | 2 | 0 | 3 | 2 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 | 1 | 3 | 2 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 1 | 2 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0 | 2 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 5 | 0 | 2 | 2 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 6 | 2 | 3 | 1 | 0 | 0
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 4 | 1 | 2 | 0 | 0 | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 19 | 1 | 5 | 7 | 1 | 5
Rash (Skin and subcutaneous tissue disorders) | 5 | 1 | 2 | 1 | 0 | 1
Hypertension (Vascular disorders) | 28 | 3 | 7 | 11 | 2 | 5
Lymphopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1 | 0 | 0
Polycythaemia (Blood and lymphatic system disorders) | 1 | 0 | 1 | 0 | 0 | 0
Angina pectoris (Cardiac disorders) | 1 | 0 | 0 | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 1
Bradycardia (Cardiac disorders) | 1 | 0 | 1 | 0 | 0 | 0
Hypertensive heart disease (Cardiac disorders) | 1 | 1 | 0 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 1 | 0 | 0 | 1 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 1
Ear pain (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 0 | 0 | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 2 | 1 | 0 | 1 | 0 | 0
Thyroid disorder (Endocrine disorders) | 1 | 0 | 0 | 1 | 0 | 0
Thyroid mass (Endocrine disorders) | 1 | 0 | 0 | 1 | 0 | 0
Cataract (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 1
Lacrimation increased (Eye disorders) | 2 | 0 | 1 | 1 | 0 | 0
Retinal vein occlusion (Eye disorders) | 2 | 0 | 0 | 1 | 0 | 1
Vision blurred (Eye disorders) | 2 | 0 | 0 | 1 | 0 | 1
Visual impairment (Eye disorders) | 1 | 0 | 0 | 0 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0
Angular cheilitis (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0
Colitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 1
Dry mouth (Gastrointestinal disorders) | 2 | 1 | 1 | 0 | 0 | 0
Duodenal ulcer (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0
Flatulence (Gastrointestinal disorders) | 2 | 0 | 1 | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 2 | 0 | 0 | 2 | 0 | 0
Gastrointestinal motility disorder (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0
Gastrointestinal tract irritation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 1
Gingival swelling (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0
Glossitis (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0
Glossodynia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 1
Haematemesis (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0
Melaena (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0
Oral pain (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 1 | 1
Pancreatitis (Gastrointestinal disorders) | 2 | 0 | 0 | 1 | 0 | 1
Periodontal disease (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0
Tooth loss (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0
Chest discomfort (General disorders) | 1 | 0 | 1 | 0 | 0 | 0
Facial pain (General disorders) | 1 | 0 | 1 | 0 | 0 | 0
Hernia (General disorders) | 1 | 0 | 0 | 0 | 0 | 1
Impaired healing (General disorders) | 1 | 0 | 0 | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 2 | 0 | 0 | 1 | 1 | 0
Pain (General disorders) | 2 | 1 | 0 | 1 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 1 | 0 | 0 | 0
Cholestasis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 2 | 0 | 0 | 2 | 0 | 0
Cystitis (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0
Erysipelas (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0
Folliculitis (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1
Helicobacter infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1
Herpes zoster (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0
Influenza (Infections and infestations) | 2 | 0 | 0 | 1 | 0 | 1
Liver abscess (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0
Otitis media (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0
Perichondritis (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1
Tinea pedis (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 2 | 1 | 0 | 0 | 1 | 0
Sunburn (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0 | 1 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0 | 1 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 0 | 1 | 0 | 0 | 0
Blood magnesium decreased (Investigations) | 1 | 0 | 1 | 0 | 0 | 0
Blood potassium decreased (Investigations) | 2 | 0 | 1 | 0 | 0 | 1
Blood triglycerides increased (Investigations) | 1 | 0 | 0 | 1 | 0 | 0
Carbon dioxide increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 1
Chest X-ray abnormal (Investigations) | 1 | 1 | 0 | 0 | 0 | 0
Haematocrit increased (Investigations) | 1 | 0 | 1 | 0 | 0 | 0
Haemoglobin decreased (Investigations) | 1 | 0 | 0 | 1 | 0 | 0
Heart rate increased (Investigations) | 1 | 0 | 0 | 1 | 0 | 0
International normalised ratio increased (Investigations) | 1 | 0 | 1 | 0 | 0 | 0
Prostatic specific antigen increased (Investigations) | 1 | 0 | 0 | 0 | 1 | 0
Troponin increased (Investigations) | 1 | 0 | 1 | 0 | 0 | 0
Urine protein/creatinine ratio increased (Investigations) | 1 | 1 | 0 | 0 | 0 | 0
White blood cell count (Investigations) | 1 | 0 | 0 | 1 | 0 | 0
White blood cell count decreased (Investigations) | 1 | 0 | 0 | 1 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 2 | 0 | 1 | 1 | 0 | 0
Glucose tolerance impaired (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 1
Gout (Metabolism and nutrition disorders) | 2 | 1 | 1 | 0 | 0 | 0
Hyperamylasaemia (Metabolism and nutrition disorders) | 2 | 1 | 0 | 1 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 1 | 1 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 2 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 1
Hyperlipidaemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 2 | 0 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 0 | 0
Hypochloraemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 0 | 0
Hypocholesterolaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 0 | 0
Polydipsia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 0 | 0
Coccydynia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1 | 1 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1 | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0
Vertebral osteophyte (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1 | 0 | 0
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 1 | 0 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 1
Aphasia (Nervous system disorders) | 1 | 0 | 1 | 0 | 0 | 0
Carotid artery thrombosis (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 1
Dysgeusia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 1
Hyperaesthesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 1
Memory impairment (Nervous system disorders) | 1 | 0 | 0 | 0 | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0 | 0 | 1 | 0 | 0
Radiculopathy (Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 1 | 0 | 1 | 0 | 0 | 0
Depression (Psychiatric disorders) | 2 | 0 | 1 | 1 | 0 | 0
Mood altered (Psychiatric disorders) | 1 | 0 | 0 | 1 | 0 | 0
Chromaturia (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 1 | 0
Chronic kidney disease (Renal and urinary disorders) | 1 | 1 | 0 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 2 | 0 | 0 | 1 | 0 | 1
Renal impairment (Renal and urinary disorders) | 1 | 0 | 0 | 1 | 0 | 0
Urethral disorder (Renal and urinary disorders) | 1 | 0 | 0 | 1 | 0 | 0
Urinary hesitation (Renal and urinary disorders) | 1 | 0 | 1 | 0 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 1 | 0 | 0 | 0 | 0
Prostatomegaly (Reproductive system and breast disorders) | 1 | 0 | 0 | 1 | 0 | 0
Pruritus genital (Reproductive system and breast disorders) | 1 | 0 | 0 | 1 | 0 | 0
Uterine haemorrhage (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0 | 0
Rales (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1 | 0
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0 | 0
Stridor (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0 | 0
Actinic keratosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0
Dermatitis psoriasiform (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 | 0 | 1 | 0 | 0 | 1
Nail disorder (Skin and subcutaneous tissue disorders) | 2 | 0 | 1 | 1 | 0 | 0
Nail dystrophy (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0
Rosacea (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0
Scab (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 1 | 0 | 1
Coronary arterial stent insertion (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 1 | 0
Tooth extraction (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 0 | 1
Peripheral arterial occlusive disease (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 1
Peripheral vascular disorder (Vascular disorders) | 1 | 1 | 0 | 0 | 0 | 0
Raynaud's phenomenon (Vascular disorders) | 1 | 0 | 0 | 1 | 0 | 0
Venous occlusion (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-11-08): https://cdn.clinicaltrials.gov/large-docs/19/NCT00828919/Prot_SAP_000.pdf